CLINICAL TRIAL: NCT04068493
Title: Enhanced Project Health: A Dissonance-Based Intervention for Obesity in Young Adults
Brief Title: A Dissonance-Based Obesity Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator is transitioning to a new faculty position at another institution.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sylvia Herbozo, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0892
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blind to the condition that participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dissonance-based obesity intervention (Experimental): Participants in this arm will receive Enhanced Project Health.
  Interventions: Behavioral: Enhanced Project Health
- Assessment Only (No Intervention): Participants in this arm will only complete the baseline assessment and 2 month assessment. They will not receive Enhanced Project Health.

INTERVENTIONS:
Behavioral: Enhanced Project Health — A dissonance-based obesity intervention consisting of eight weekly groups sessions (1.5 hours).
  Arms: Dissonance-based obesity intervention

SUMMARY:
This project will examine the feasibility and acceptability of Enhanced Project Health, a dissonance-based obesity intervention, and whether this intervention results in significantly greater reductions in weight and improvements in lifestyle behaviors than an assessment only condition. Participants will be young adults enrolled in college.

DETAILED DESCRIPTION:
Approximately 34% of college students are overweight/obese. However, few behavioral weight loss (BWL) interventions have been developed for young adults in college. Research suggests that standard BWL interventions are not addressing the needs of young adults as they have shown poorer retention rates and weight loss compared to older adults in BWL trials. Standard BWL interventions are also time-intensive and are not conducive to inexpensive dissemination.

The primary aim of this project is to examine the feasibility and acceptability of Enhanced Project Health, a dissonance-based obesity intervention for young adults enrolled in college. Enhanced Project Health is based on Project Health, a dissonance-based obesity prevention program, which has been shown to significantly decrease weight gain and future overweight/obesity onset compared to a matched intervention and minimal intervention control condition in young adults. The current intervention was expanded to consist of eight weekly group sessions and to address sleep, in addition to diet and physical activity. The secondary aim is to test the hypothesis that Enhanced Project Health will result in significantly greater reductions in weight and improvements in lifestyle behaviors compared to an assessment only condition.

ELIGIBILITY:
Inclusion Criteria:

1. Young adults of ages 18 to 25.
2. Enrolled as a college student.
3. Body mass index of 25 or more (overweight/obese) based on measured height and weight.

Exclusion Criteria:

1. Diagnosis of bulimia nervosa according to DSM-5 criteria.
2. Diagnosis of obstructive sleep apnea.
3. Participation in interventions for weight loss or disordered eating behaviors.
4. Current use of prescription drugs for weight loss or disordered eating behaviors.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible young adults that agree to participate in the study | Up to 1 month
  This will be defined as a percentage of young adults that agree to participate in study out of the young adults screened for the study.
Time for recruitment | Up to 1 month
  This will be defined as time (weeks and days) from initial contact with research staff to randomization into the study.
Attendance rate of participants | Assessed at 2 months
  This will be defined as the percentage of participants attending 75% of the group sessions.
Retention rate of participants | Assessed at 2 months
  This will be defined as the percentage of participants remaining in the study at the post-intervention assessment.
Program Evaluation Questionnaire - Each Group Session | Assessed from week 1 to week 8
  This questionnaire was developed for this study. It will assess the acceptability of the intervention and will be administered at the end of each group session. Participants will be asked to rate the usefulness of the session on one item with a scale ranging from 1 to 5. Total scores range from 1 to 5. Higher scores indicate more usefulness.
  Participants will also be asked to respond to open-ended questions about each group session. These questions will assess the most favorable aspects, least favorable aspects, and areas of improvements. Responses will be coded using a variation of the long table approach emphasizing frequency, specificity, emotion, and extensiveness. Codes will be examined to identify themes.
Program Evaluation Questionnaire - Overall Program | Assessed at week 8
  This questionnaire was developed for this study. It will assess the program with regard to effectiveness and satisfaction as well as characteristics of the group leaders (clarity, knowledge, experience, respect) using a scale ranging from 1 to 5. Total scores range from 8 to 40. Higher scores indicate more favorable responses. This questionnaire will be administered at the end of the last group session.

SECONDARY OUTCOMES:
Body Mass Index (kg/m^2) | Baseline to 2 months
  Body Mass Index will be calculated using measured weight and height (kg/m^2)
International Physical Activity Questionnaire-Short Form (IPAQ-S) | Baseline to 2 months
  The International Physical Activity Questionnaire-Short Form will assess walking, moderate-intensity activity, and vigorous-intensity activity. The scores for each type of physical activity are converted to MET-minutes/week as defined by the following: Walking MET-minutes/week = 3.3 * walking minutes * walking days; Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days; Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days; Total physical activity MET-minutes/week = sum of Walking + Moderate + Vigorous MET-minutes/week scores. The total score will be computed by summing the duration (in minutes) and frequency (days) of each activity. Higher duration and frequency indicate more engagement in physical activity. The pattern of physical activity can also be classified as low, moderate, or high based on the total score.
Actigraph GT3XP-BTLE | Baseline to 2 months
  An accelerometer will record physical activity for a 1 week period
Pittsburgh Sleep Quality Index (PSQI) | Baseline to 2 months
  The Pittsburgh Sleep Quality Index will assess the quality and patterns of sleep using a scale ranging from 0 to 3. Total scores range from 8 to 57. Higher scores indicate greater sleep disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Herbozo, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Neuropsychiatric Institute, University of Illinoist at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No